CLINICAL TRIAL: NCT03479905
Title: A Prospective, Randomized Trial Comparing the Use of High Flow Nasal Cannula, Standard Face Mask and Standard Nasal Cannula in Morbidly Obese Patients With High Risk of Obstructive Sleep Apnea Undergoing Colonoscopy
Brief Title: The Use of High Flow Nasal Cannula, Standard Face Mask and Standard Nasal Cannula in Morbidly Obese Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemia
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christina Riccio, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 102017-005
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Desaturation of Blood; Colonoscopy
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Salter nasal cannula (Sham Comparator): A Salter nasal cannula will be used at 4L/ minute during the colonoscopy. The FiO2 delivered to the patient at this rate has been shown to be equal to 36%
  Interventions: Other: Salter nasal cannula
- Face mask group (Sham Comparator): A standard face mask will be used at 8L/minute during the colonoscopy. The FiO2 delivered to the patient at this rate has been shown to be equal to 60%.
  Interventions: Other: Face mask
- High Flow Oxygen delivery (Experimental): Oxygen will be delivered by using high flow nasal cannula
  Interventions: Device: High Flow Nasal Cannula

INTERVENTIONS:
Other: Salter nasal cannula — Oxygen will be delivered via standard nasal cannula during colonoscopy
  Arms: Salter nasal cannula
Other: Face mask — Oxygen will be delivered via face mask during colonoscopy
  Other Names: Standard Face Mask
  Arms: Face mask group
Device: High Flow Nasal Cannula — A high flow nasal cannula will be placed on the patient at a setting of FiO2 100% and titrated up to 60L/min depending on patient tolerance. 60 L/min is the max flow rate and will be used as tolerated for maximum benefit.
  Other Names: Device The Comfort Flo system
  Arms: High Flow Oxygen delivery

SUMMARY:
It is standard practice in the United States and many parts of world to perform Gastrointestinal endoscopy with the patient under deep intravenous sedation. Obesity is accepted as a patient specific risk factor for hypoxic events during procedural sedation for GI endoscopic procedures. The obese population has a higher prevalence of obstructive sleep apnea (OSA), which is characterized by repeated obstruction of the upper airway, and leads to apnea and desaturation. This prospective, randomized study was designed to compare the effectiveness of the high flow nasal cannula, standard nasal cannula and standard face mask in morbidly obese patients with a high risk of sleep apnea, (BMI greater than 40, STOPBANG greater or equal to 5) receiving deep intravenous sedation during colonoscopies. This study will assess which method leads to a lower incidence of intraoperative desaturation events compared to the current standard of care.

DETAILED DESCRIPTION:
The prevalence of morbid obesity is increasing worldwide. As the severity of obesity increases, the incidence of diagnosed obstructive sleep apnea also rises. Studies have shown an incidence of sleep apnea as high as 64% in patients with a body mass index (BMI) over 40 and 100% in patients with a BMI greater than 60. Patients with OSA have been shown to have significant desaturations under intravenous sedation due to airway narrowing and obstruction. Several studies have also shown that morbidly obese subjects, independent of a diagnosis of OSA, run a higher perioperative risk of adverse airway events, including hypoxia. Providing anesthesia for this patient population is challenging and requires careful titration of drugs and superb airway management skills.

The current standard of care for oxygen delivery in this setting is a Salter nasal cannula. Humidified high flow nasal cannula (HFNC) oxygen therapy utilizes an air oxygen blend allowing from 21% to 100% FiO2 delivery and generates up to 60 L/min flow rates. The gas is heated (35 to 40 degree Celsius) and humidified through an active heated humidifier and delivered via a single limb heated inspiratory circuit (to avoid heat loss and condensation) to the subject through a large diameter nasal cannula. Theoretically, HFNC offers significant advantages in oxygenation and ventilation over conventional methods. Constant high flow oxygen delivery provides steady inspired oxygen fraction (FiO2) and decreases oxygen dilution. It also washes out physiologic dead space and generates positive end expiration pressure (PEEP) that augments ventilation.

Some studies have demonstrated a positive effect of HFNC on the apnea-hypopnea index (AHI) showing that use of HFNC could decrease hypoxic episodes in subjects with repetitive upper airway obstruction such as obstructive sleep apnea. The STOP-BANG questionnaire (SB) has been used successfully to screen patients undergoing therapeutic endoscopic procedures at higher risk for sedation-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80
* Subjects undergoing colonoscopies
* Morbidly obese BMI equal or greater than 40
* STOPBANG score equal or greater than 5

Exclusion Criteria:

* Subjects deemed hemodynamically unstable by the anesthesia team
* Subjects who are an aspiration risk and will require endotracheal intubation.
* Pregnancy
* Subjects with an allergy to propofol
* Patients who are unable to tolerate the high flow nasal cannula secondary to discomfort
* Subjects unwilling to sign consent
* Patients that received medications other than lidocaine and propofol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Riccio, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Helath Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Salter Nasal Cannula: A Salter nasal cannula will be used at 4L/ minute during the colonoscopy. The FiO2 delivered to the patient at this rate has been shown to be equal to 36%
  Salter nasal cannula: Oxygen will be delivered by using standard nasal cannula
Period: Overall Study
Arm/Group | Salter Nasal Cannula | Face Mask Group | High Flow Oxygen Delivery
Started | 47 | 48 | 48
Completed | 43 | 43 | 43
Not Completed | 4 | 5 | 5
Not completed — Other airway method used | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salter Nasal Cannula | Face Mask Group | High Flow Oxygen Delivery | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.55 (8.10) | 58.23 (6.73) | 57.55 (10.04) | 57.44 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 28 | 87
  Male | 15 | 12 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 10 | 33
  Not Hispanic or Latino | 30 | 31 | 32 | 93
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 22 | 19 | 62
  White | 20 | 21 | 23 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 43 | 129
Stop Bang Score [Median (Inter-Quartile Range); unit: Stop Bang Score on a scale of 0 to 8] — Stop Bang Score for Obstructive Sleep Apnea on a scale of 0 to 8. A score of 2 or less is considered low risk, and a score of 5 or more is high risk for having either moderate or severe Obstructive Sleep Apnea.
  Stop Bang Score on a scale of 0 to 8 | 6 [6 to 7] | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7]
Preoperative oxygen saturation (SpO2) [Median (Inter-Quartile Range); unit: Percentage of oxygen saturation] | 97.5 [96 to 98] | 98 [96 to 99] | 97 [96 to 98] | 98 [96 to 98]

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2 )
Description: The frequency of desaturation episodes (SpO2 <90%)
Time Frame: Intraoperative period, an average of 1 hour
Measure: Median (Inter-Quartile Range); unit: Desaturation episodes
Arm/Group | Salter Nasal Cannula | Face Mask Group | High Flow Oxygen Delivery
Number analyzed (Participants) | 43 | 43 | 43
Desaturation episodes | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Salter Nasal Cannula vs Face Mask Group vs High Flow Oxygen Delivery; Test type: Superiority; p = 0.0004, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: During hospital stay, an average of 6 hours
Arm/Group | Salter Nasal Cannula | Face Mask Group | High Flow Oxygen Delivery
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03479905/Prot_SAP_ICF_001.pdf